CLINICAL TRIAL: NCT06979921
Title: Breast Cancer Early-stage Detection by Liquid Biopsy in Peripheral Blood: a Retrospective and Prospective Study
Brief Title: PERformance of Multi-Cancer Early-detectIon Based on Various Biomarkers in fEmale BREAST Cancers, PERCEIVE-BREAST
Status: Active, not recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Guangzhou Bruning Rock Bioengineering Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: JSSRM-2021013
Record Dates: First submitted 2022-05-29; First posted 2025-05-20 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-04

CONDITIONS: Cancer
Keywords: cancer; liquid biopsy; early detection; cell-free DNA methylation
MeSH Terms: conditions — Neoplasms | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer arm: Baseline blood samples will be collected from participants with new diagnosis breast cancer.
  Interventions: Device: Blood test
- Benign disease arm: Baseline blood samples will be collected from participants with new diagnosis breast benign disease.
  Interventions: Device: Blood test

INTERVENTIONS:
Device: Blood test — Blood test

SUMMARY:
This study is a retrospective and prospective study aimed to develop and validate the performance of multi-omics assays for early detection of female breast cancer. The study will enroll approximately 496 participants including participants with breast cancers and participants with breast benign diseases.

ELIGIBILITY:
Inclusion Criteria for All Participants:

* Able to provide a written informed consent.
* Female, at least 18 years old.

Additional Inclusion Criteria for Breast Cancer Participants:

* Pathologically confirmed breast cancer diagnosis or highly suspicious for breast cancer within 42 days prior to blood draw.
* No prior cancer treatment before the blood draw.

Additional Inclusion Criteria for Breast Benign Disease Participants:

* Pathologically confirmed breast cancer diagnosis or highly suspicious of breast benign diseases within 90 days prior to blood draw.
* No prior radical treatment before the blood draw.

Exclusion Criteria for All Participants:

* During pregnancy or lactation.
* Recipient of organ transplant or prior non-autologous (allogeneic) bone marrow or stem cell transplant.
* Recipient of blood transfusion within 7 days prior to blood draw.
* Recipient of anti-tumor drugs to treat non-cancer diseases prior to blood draw, such as rheumatic drugs (methotrexate, cyclophosphamide, or azathioprine), or endocrine drugs (tamoxifen).

Additional Exclusion Criteria for Breast Cancer Participants:

* Multiple primary tumors.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible participants will be recruited from medical centers and assigned into two arms, including participants with new diagnosis of breast cancer or breast benign disease.
Sampling Method: Non-Probability Sample
Enrollment: 496 (Actual)
Dates: Start 2021-07-10 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of cell-free DNA (cfDNA) methylation in the detection of breast cancer. | 48 months
The sensitivity and specificity of circulating tumor DNA (ctDNA) mutations in the detection of breast cancer. | 48 months
The sensitivity and specificity of blood miRNA in the detection of breast cancer. | 48 months

SECONDARY OUTCOMES:
The sensitivity and specificity of the multi-omics model in the detection of breast cancer. | 48 months
The sensitivity and specificity of various omics-based models for detecting different molecular subtypes of breast cancer. | 48 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Jiangsu Provincial People's Hospital, Nanjing, Jiangsu
  - The Affiliated Hospital of Medical College Qingdao University, Qingdao, Shandong